CLINICAL TRIAL: NCT03239769
Title: A Study to Evaluate and Compare the Surgical Outcomes, Aesthetic Effects and Incision Length of Different Access Procedures in Patients With DTC
Brief Title: Compare the Aesthetic Effect of Different Thyroidectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Xiao Ma, Associate chief physician, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XMa-001
Record Dates: First submitted 2017-08-01; First posted 2017-08-04 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Differentiated Thyroid Carcinoma (DTC)
Keywords: Thyroid surgery; Thyroidectomy; Minimally invasive access; Aesthetic principle; POSAS
MeSH Terms: interventions — Thyroidectomy

STUDY DESIGN:
Intervention Model Description: These patients were individually randomly assigned (1:1:1 ratio) into the conventional access group (CA), the aesthetic principles access group (APA) or the minimally invasive access group (MIA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional access group (CA) (Active Comparator): A 4- to 5-cm incision was created, subplatysmal flaps were raised, and the strap muscles were mobilized. Then, the superior pole of the thyroid gland was exposed and the gland was delivered through the surgical incision, and the thyroid isthmus was divided. Finally, CLND was performed. The strap muscles were re-approximated with No.1 silk suture. The full-thickness skin was closed with interrupted monofilament.
  Interventions: Procedure: thyroidectomy
- aesthetic principles access group (APA) (Experimental): The key difference focused on the disposal incision using aesthetic principles, which are depicted below. The incision was protected by Vaseline ointment. Excessive skin traction was avoided to prevent the injury on the skin edge. Bleeding was stanched with a low-power bipolar coagulation device. The surgical field does not have to be pulled in every direction to show the full operation field. The cervical linea alba was closed by continuous sutures with 3-0 absorbable Vicryl sutures. Interrupted sutures of 4-0 Vicryl were used to re-approximate the subcutaneous tissues. The epidermis was fixed with 3M steri-strip elastic skin closures rather than skin sutures.
  Interventions: Procedure: thyroidectomy
- minimally invasive access group (MIA) (Experimental): With the MIA approach, a shorter incision of between 3 and 4 cm was created. The procedure used the Harmonic scalpel as an auxiliary device. First, the isthmus was divided. Second, the lower pole of the thyroid was dissected from the adipose tissue, and the inferior thyroid vessels were divided close to the thyroid gland for mobilization. The RLN and parathyroid glands were carefully dissected. Third, the superior pole of the thyroid gland was disconnected. Finally, CLND was performed. The closure procedure for the incision was similar to that for APA.
  Interventions: Procedure: thyroidectomy

INTERVENTIONS:
Procedure: thyroidectomy — Thyroidectomies have different approaches. The aim of this study was to evaluate and compare the aesthetic effects of different access procedures in patients with differentiated thyroid carcinoma (DTC).

SUMMARY:
One hundred twenty female patients who underwent thyroidectomy were evenly distributed into three groups: conventional access (CA), aesthetic principles access (APA) and minimally invasive access (MIA). The Patient and Observer Scar Assessment Scale (POSAS) was used as the assessment tool for the linear scar. After one year follow-up, the cosmetic outcomes were assessed.

DETAILED DESCRIPTION:
A prospective study in patients with DTC at the Department of Head and Neck Surgery at Perking University Cancer Hospital (also called Beijing Cancer hospital). A total of 120 female patients who underwent surgical treatment for DTC were enrolled in the study from June 2012 to June 2014. All patients were diagnosed with DTC through preoperative fine needle aspiration biopsy pathology. These patients were individually randomly assigned (1:1:1 ratio) into the conventional access group (CA), the aesthetic principles access group (APA) or the minimally invasive access group (MIA). Lobectomy plus ipsilateral central lymph node dissection (CLND) was adopted in each patient. DTC staging was T1N0M0 or T1N1M0. The investigators retrieved the patients' information, including age, incision length, incision closure procedure, incidence of complications, and cosmetic assessment from patients' medical records. Patients with other medical diseases, such as diabetes or obesity, a smoking history, a keloid tendency, a history of radiotherapy to the head and neck, or with incomplete information, were excluded. RLN function was evaluated by electronic fiber laryngoscopy 6 months postoperatively. The follow-up time was 12.3 months. The research was reviewed and approved by the Ethics Committee of Peking University Cancer Hospital, and informed consent was obtained from all patients to publish the information/image(s) in an online open-access publication. The study was open-label with no blinding of patients, clinicians, or research staff.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with DTC through preoperative fine needle aspiration biopsy pathology.
* DTC staging was T1N0M0 or T1N1M0.
* Female
* Age over 18 years
* Subjects who fully understand the study process, participate voluntarily

Exclusion Criteria:

* Patients with other medical diseases, such as diabetes or obesity, a smoking history, a keloid tendency, a history of radiotherapy to the head and neck, or with incomplete information.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) | 12 months post-operation
  The POSAS scale is a reliable and feasible tool for linear scar evaluation. The POSAS included the observer scale and the patient scale. The Observer Scar Assessment Scale (OSAS) score was obtained by the same observer; this scale includes 5 items graded on a 10-point scale with 1 indicating normal skin and 10 indicating the worst scar imaginable. A summary score of 5 indicates normal skin, and a summary score of 50 is the worst possible scar result. The Patient Scar Assessment Scale (PSAS) consists of 6 items. All items are graded by the patient on a 10-point scale; a summary score of 6 to 60 represents the range from normal skin to the worst imaginable scar. After scoring the items, the observer and the patients rated the overall scar appearance on a visual analogue scale corresponding to a 10-point scale.

SECONDARY OUTCOMES:
Scar length | 12 months post-operation
  Using ruler to measure the length of the scar, accuracy to millimeter
Operation time | Day 1 (on the day of operation)
  From incision to suture completed (record the duration from start of operation to the end of operation)
Blood loss | Day 1 (on the day of operation)
  Blood loss from incision to suture completed (record the blood loss from start of operation to the end of operation)
Amount of drainage | till extubation, an average of 48 hours post-operation
  Record the amount of the drainage from end of surgical procedure to extubation of drainage
Duration of drainage | till extubation, an average of 48 hours post-operation
  Record the duration (days) of the drainage, from end of surgical procedure to extubation of drainage
Number of CLND | up to 2 weeks post-operation
  Record the number of central lymph nodes

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Ma, Doctor, Principal Investigator — Peking University Cancer Hospital & Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma X, Xia QJ, Li G, Wang TX, Li Q. Aesthetic principles access thyroidectomy produces the best cosmetic outcomes as assessed using the patient and observer scar assessment scale. BMC Cancer. 2017 Sep 18;17(1):654. doi: 10.1186/s12885-017-3645-2. PMID 28923027